CLINICAL TRIAL: NCT01636154
Title: Clinical Application and Basic Study of Medicinal Fractions-based Herbal Combinations:A Prospective Randomized Controlled Multi-site Clinical Trial About Fractions-based Herbal Combinations of Clearing Heat and Promoting Blood Circulation
Brief Title: Clinical Application and Basic Study of Medicinal Fractions-based Herbal Combinations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yunling Zhang (Other)
Collaborators: Shandong University of Traditional Chinese Medicine (Other); Huairou Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor-Investigator, Yunling Zhang, President of of Dongfang Hospital, Dongfang Hospital Beijing University of Chinese Medicine
Organization: Dongfang Hospital Beijing University of Chinese Medicine (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: BUCMDFH9634
Record Dates: First submitted 2012-06-29; First posted 2012-07-10 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Ischemic Stroke
Keywords: fire-heat syndrome; blood stasis syndrome; method of clearing heat; method of promoting blood circulation; medicinal fractions-based herbal combinations
MeSH Terms: conditions — Ischemic Stroke | interventions — Panax notoginseng extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- The basic treatment (No Intervention): Comply to the Chinese guidelines of acute ischemic stroke in 2010
- Clearing heat (Other): Treat with KDZ injection on the basis of the basic treatment
  Interventions: Drug: Ixeris of sonchifolia Hance
- Promoting blood circulation (Other): Treat with Xueshuantong injection on the basis of the basic treatment
  Interventions: Drug: Panax notoginseng saponins
- Clearing heat & Promoting blood circulation (Experimental): Treat with both KDZ injection and Xueshuantong injection on the basis of the basic treatment
  Interventions: Drug: Ixeris of sonchifolia Hance combined with Panax notoginseng saponins

INTERVENTIONS:
Drug: Ixeris of sonchifolia Hance — KDZ40ml+0.9%N.S.250ml,ivdrip,qd of each 14-day cycle.Number of cycles:one.
  Other Names: KDZ injection
  Arms: Clearing heat
Drug: Panax notoginseng saponins — Xueshuantong450mg+0.9%N.S.250ml,ivdrip,qd of each 14-day cycle.Number of cycles:one.
  Other Names: Xueshuantong injection
  Arms: Promoting blood circulation
Drug: Ixeris of sonchifolia Hance combined with Panax notoginseng saponins — KDZ40ml+0.9%N.S.250ml,ivdrip;0.9%N.S.50ml,ivdrip;Xueshuantong450mg+0.9%N.S.250ml,ivdrip.qd of each 14-day cycle.Number of cycles:one.
  Arms: Clearing heat & Promoting blood circulation

SUMMARY:
The purpose of this study is to investigate the efficacy of fractions-based herbal combinations of clearing heat and promoting blood circulation treating acute ischemic stroke and the potential mechanism of it.

DETAILED DESCRIPTION:
The interaction between fire-heat and blood stasis is a significant mechanism underlying pathogenesis and progress in acute ischemic stroke according to TCM theory.Clinical therapeutic effects are achieved with wide application of Ixeris of sonchifolia Hance components (KDZ injection) representing method of clearing heat and Panax notoginseng saponins components (Xueshuantong injection) representing method of promoting blood circulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute ischemic stroke
* Patients with fire-heat syndrome
* Stoke onset within 48 hours
* NIHSS scores range from 5 points to 25 points
* Age from forty to seventy-five,gender not limited
* Informed and signed the consent

Exclusion Criteria:

* Cardiogenic cerebral embolism,stroke caused by other reasons or the unexplained
* Patients suitable for thrombolytic therapy(rt-PA, urokinase)
* Patients have received thrombolytic therapy
* Patients with serious diseases of heart,lungs,liver,kidneys
* Patients with bleeding or bleeding tendency recently
* Pregnant or lactating women
* Pre-existing neurological or psychiatric diseases that could confound the study results
* Patients be allergic to alcohol,Ixeris of sonchifolia Hance components (KDZ injection) or Panax notoginseng saponins components (Xueshuantong injection)
* Patients have participated in other clinical trials within 3 months

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-01; Primary Completion 2016-03 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yunling Zhang, PhD,MD, Study Chair — Dongfang Hospital Beijing University of Chinese Medicine
Locations (3):
- China (3):
  - Department of Neurology,Dongfang Hospital,Beijing University of Chinese Medicine, Beijing, Beijing Municipality
  - Department of Neurology,Huairou Hospital of Traditional Chinese Medicine, Beijing, Beijing Municipality
  - Department of Neurology,Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Jinan, Shandong

REFERENCES:
- [Derived] Liu X, Jin X, Chen B, Liu X, Liang X, Fang X, Wu H, Fu X, Zheng H, Ding X, Duan N, Zhang Y. Effects of Kudiezi Injection on Serum Inflammatory Biomarkers in Patients with Acute Cerebral Infarction. Dis Markers. 2018 Sep 2;2018:7936736. doi: 10.1155/2018/7936736. eCollection 2018. PMID 30245755